CLINICAL TRIAL: NCT03614702
Title: Safety and Immunogenicity Evaluation of Different Sequential Immunization Schedules of Type1+2 Bivalent Oral Poliovirus Vaccine(bOPV) Co-administered With Inactived Poliovirus Vaccine(IPV) in Infants Aged 2 Months: a Randomized, Double Blind, Single Center, Parallel Trial
Brief Title: Clinic Trial to Evaluate the Safety and Immunogenicity by Different Sequential Schedules of bOPV and IPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: bOPV-PRO-001
Record Dates: First submitted 2017-03-03; First posted 2018-08-03 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Poliomyelitis
Keywords: bOPV; IPV; sequential immunization; immunogenecity; safety
MeSH Terms: conditions — Poliomyelitis | interventions — Candy; Poliovirus Vaccine, Oral; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (12):
- 1-dose cIPV + 2-doses bOPV (Candy) (Experimental): cIPV: Inactivated Poliomyelitis Vaccine Made from Wild Polio Strains Produced by Sanofi Pasteur Co., Ltd. 0.5ml/dose
  bOPV (Candy): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences . 1g/pill,10 pills/pach,one pill each time; each pill containing polio virus≥5.92 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 3 polio virus ≥5.3lgCCID50.
  Interventions: Biological: 1-dose cIPV + 2-doses bOPV (Candy)
- 1-dose sIPV + 2-doses bOPV (Candy) (Experimental): sIPV: Inactivated Poliomyelitis Vaccine Made from Sabin Strains Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences 0.5ml/dose
  bOPV (Candy): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 1g/pill,10 pills/pach,one pill each time;each pill containing polio virus≥5.92 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 3 polio virus ≥5.3lgCCID50.
  Interventions: Biological: 1-dose sIPV + 2-doses bOPV (Candy)
- 2-doses cIPV + 1-dose bOPV (Candy) (Experimental): cIPV: Inactivated Poliomyelitis Vaccine Made from Wild Polio Strains Produced by Sanofi Pasteur Co., Ltd. 0.5ml/dose
  bOPV (Candy): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 1g/pill,10 pills/pach,one pill each time; each pill containing polio virus≥5.92 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 3 polio virus ≥5.3lgCCID50
  Interventions: Biological: 2-doses cIPV + 1-dose bOPV (Candy)
- 2-doses sIPV + 1-dose bOPV (Candy) (Experimental): sIPV: Inactivated Poliomyelitis Vaccine Made from Sabin Strains Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml/dose
  bOPV (Candy): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 1g/pill,10 pills/pach,one pill each time; each pill containing polio virus≥5.92 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 3 polio virus ≥5.3lgCCID50
  Interventions: Biological: 2-doses sIPV + 1-dose bOPV (Candy)
- 2-doses cIPV + 1-dose tOPV (Candy) (Experimental): cIPV: Inactivated Poliomyelitis Vaccine（Vero） Made from Wild Polio Strains Produced by Sanofi Pasteur Co., Ltd. 0.5ml/dose
  tOPV (Candy): Trivalent oral attenuated live poliomyelitis vaccine against type 1, type 2 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Beijing Tiantan Biological Products Co., Ltd. 1g/pill,10 pills/pach;each pill containing polio virus≥5.95 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 2 polio virus ≥4.8lgCCID50，type 3 polio virus ≥5.3lgCCID50
  Interventions: Biological: 2-doses cIPV + 1-dose tOPV (Candy)
- 2-doses sIPV + 1-dose tOPV (Candy) (Experimental): sIPV: Inactivated Poliomyelitis Vaccine Made from Sabin Strains Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences 0.5ml/dose
  tOPV (Candy): Trivalent oral attenuated live poliomyelitis vaccine against type 1, type 2 and type 3 in Dragee Candy (Human Diploid Cell) Produced by Beijing Tiantan Biological Products Co., Ltd.1g/pill,10 pills/pach,one pills each time;each pill containing polio virus≥5.95 lgCCID50 including type1 polio virus≥5.8 lgCCID50，type 2 polio virus ≥4.8lgCCID50，type 3 polio virus ≥5.3lgCCID50
  Interventions: Biological: 2-doses sIPV + 1-dose tOPV (Candy)
- 1-dose cIPV + 2-doses bOPV (Liquid) (Experimental): cIPV: Inactivated Poliomyelitis Vaccine（Vero） Made from Wild Polio Strains Produced by Sanofi Pasteur Co., Ltd. 0.5ml/dose
  bOPV (Liquid): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml or 1.0ml each bottle;total content of polio virus≥7.12lgCCID50/ml，type1 polio virus≥7.0 lgCCID50/ml，type 3 polio virus ≥6.5lgCCID50/ml.(2 drops per person;be be equivalent to 0.1ml each person )
  Interventions: Biological: 1-dose cIPV + 2-doses bOPV (Liquid)
- 1-dose sIPV + 2-doses bOPV (Liquid) (Experimental): sIPV: Inactivated Poliomyelitis Vaccine Made from Sabin Strains Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml/dose
  bOPV (Liquid): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml or 1.0ml each bottle;total content of polio virus≥7.12lgCCID50/ml，type1 polio virus≥7.0 lgCCID50/ml，type 3 polio virus ≥6.5lgCCID50/ml.(2 drops per person;be be equivalent to 0.1ml each person )
  Interventions: Biological: 1-dose sIPV + 2-doses bOPV (Liquid)
- 2-doses cIPV + 1-dose bOPV (Liquid) (Experimental): cIPV: Inactivated Poliomyelitis Vaccine Made from Wild Polio Strains Produced by Sanofi Pasteur Co., Ltd. 0.5ml/dose
  bOPV (Liquid): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml or 1.0ml each bottle;total content of polio virus≥7.12lgCCID50/ml，type1 polio virus≥7.0 lgCCID50/ml，type 3 polio virus ≥6.5lgCCID50/ml.(2 drops per person;be be equivalent to 0.1ml each person )
  Interventions: Biological: 2-doses cIPV + 1-dose bOPV (Liquid)
- 2-doses sIPV + 1-dose bOPV (Liquid) (Experimental): sIPV: Inactivated Poliomyelitis Vaccine Made from Sabin Strains Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml/dose
  bOPV (Liquid): bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3 (Human Diploid Cell) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 0.5ml or 1.0ml each bottle,total content of polio virus≥7.12lgCCID50/ml，type1 polio virus≥7.0 lgCCID50/ml，type 3 polio virus ≥6.5lgCCID50/ml.(2 drops per person;be be equivalent to 0.1ml each person )
  Interventions: Biological: 2-doses sIPV + 1-dose bOPV (Liquid)
- 2-doses cIPV + 1-dose tOPV (Liquid) (Experimental): cIPV: Inactivated Poliomyelitis Vaccine Made from Wild Polio Strains Produced by Sanofi Pasteur Co., Ltd. 0.5ml/dose
  tOPV(Liquid) Trivalent oral attenuated live poliomyelitis vaccine against type 1, type 2 and type 3 in Dragee Candy (Vero) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 1.0ml each bottle,total content of polio virus≥7.15lgCCID50/ml，type1 polio virus≥ 7.0 lgCCID50/ml，type2 polio virus ≥ 6.0lgCCID50/ml，type 3 polio virus≥ 6.5lgCCID50/ml.(2 drops per person;be be equivalent to 0.1ml each person )
  Interventions: Biological: 2-doses cIPV + 1-dose tOPV (Liquid)
- 2-doses sIPV + 1-dose tOPV (Liquid) (Experimental): sIPV: Inactivated Poliomyelitis Vaccine Made from Sabin Strains Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences.0.5ml/dose
  Trivalent oral attenuated live poliomyelitis vaccine against type 1, type 2 and type 3 in Dragee Candy (vero) Produced by Institute of Medical Biology, Chinese Academy of Medical Sciences. 1.0ml each bottle,total content of polio virus≥7.15lgCCID50/ml，type1 polio virus≥7.0 lgCCID50/ml，type 2 polio virus ≥ 6.0lgCCID50/ml，type 3 polio virus ≥ 6.5lgCCID50/ml.(2 drops per person;be be equivalent to 0.1ml each person )
  Interventions: Biological: 2-doses sIPV + 1-dose tOPV (Liquid)

INTERVENTIONS:
Biological: 1-dose cIPV + 2-doses bOPV (Candy) — Health subjects received 1-dose cIPV intramuscularly in the centre of anterolateral thigh followed by 2-doses bOPV(Candy) through mouth at 0, 28, 56 days schedule.
  Arms: 1-dose cIPV + 2-doses bOPV (Candy)
Biological: 1-dose sIPV + 2-doses bOPV (Candy) — Health subjects received 1-dose sIPV intramuscularly in the centre of anterolateral thigh followed by 2-doses bOPV(Candy) through mouth at 0, 28, 56 days schedule.
  Arms: 1-dose sIPV + 2-doses bOPV (Candy)
Biological: 2-doses cIPV + 1-dose bOPV (Candy) — Health subjects received 2-doses cIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose bOPV(Candy) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses cIPV + 1-dose bOPV (Candy)
Biological: 2-doses sIPV + 1-dose bOPV (Candy) — Health subjects received 2-doses sIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose bOPV(Candy) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses sIPV + 1-dose bOPV (Candy)
Biological: 2-doses cIPV + 1-dose tOPV (Candy) — Health subjects received 2-doses cIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose tOPV(Candy) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses cIPV + 1-dose tOPV (Candy)
Biological: 2-doses sIPV + 1-dose tOPV (Candy) — Health subjects received 2-doses sIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose tOPV(Candy) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses sIPV + 1-dose tOPV (Candy)
Biological: 1-dose cIPV + 2-doses bOPV (Liquid) — Health subjects received 1-dose cIPV intramuscularly in the centre of anterolateral thigh followed by 2-doses bOPV(Liquid) through mouth at 0, 28, 56 days schedule.
  Arms: 1-dose cIPV + 2-doses bOPV (Liquid)
Biological: 1-dose sIPV + 2-doses bOPV (Liquid) — Health subjects received 1-dose sIPV intramuscularly in the centre of anterolateral thigh followed by 2-doses bOPV(Liquid) through mouth at 0, 28, 56 days schedule.
  Arms: 1-dose sIPV + 2-doses bOPV (Liquid)
Biological: 2-doses cIPV + 1-dose bOPV (Liquid) — Health subjects received 2-doses cIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose bOPV(Liquid) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses cIPV + 1-dose bOPV (Liquid)
Biological: 2-doses sIPV + 1-dose bOPV (Liquid) — Health subjects received 2-doses sIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose bOPV(Liquid) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses sIPV + 1-dose bOPV (Liquid)
Biological: 2-doses cIPV + 1-dose tOPV (Liquid) — Health subjects received 2-doses cIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose tOPV(Liquid) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses cIPV + 1-dose tOPV (Liquid)
Biological: 2-doses sIPV + 1-dose tOPV (Liquid) — Health subjects received 2-doses sIPV intramuscularly in the centre of anterolateral thigh followed by 1-dose tOPV(Liquid) through mouth at 0, 28, 56 days schedule.
  Arms: 2-doses sIPV + 1-dose tOPV (Liquid)

SUMMARY:
With the progress of the eradication of polio, bivalent oral attenuated live poliomyelitis vaccine against type 1 and 3 (bOPV) and inactivated poliomyelitis vaccine made by Sabin strain (sIPV) are required to use in the "Strategy of Polio Eradication & Endgame Strategic Plan 2013-2018" worldwide.

To evaluate the safety and immunogenicity by different sequential schedules of bOPV/tOPV with IPV(sIPV/cIPV), a randomized, double blind, single center and parallel phase Ⅲ clinic trial was performed in Infants of two-month-old in Guangxi Province, China.

DETAILED DESCRIPTION:
According to the requirement of the Strategy of Polio Eradication & Endgame Strategic Plan 2013-2018, bivalent oral attenuated live poliomyelitis vaccine against type 1 and 3 (bOPV) and inactivated poliomyelitis vaccine made by Sabin strain (sIPV) need to be used to eradiation both the wild poliovirus and vaccine-derived poliovirus.

By studying different sequential immunization schedules of bOPV(candy/liquid) with IPV(cIPV/sIPV) to evaluate the safety and immunogenicity of bivalent oral poliomyelitis vaccine co-administered with IPV in healthy Infants. A randomized, double blind, single center and parallel phase Ⅲ clinic trial was performed in Guangxi Province in China. A total of 1200 infants at 2 months old were selected, and randomly divided into 12 different groups (100 individuals were included in each group) administrated the vaccines at 0, 28, 56 days schedule. The bOPV(bivalent oral attenuated live poliomyelitis vaccine against type 1 and type 3), tOPV(trivalent OPV against type 1, type 2 and type 3), sIPV (Inactivated Poliomyelitis Vaccine Made from Sabin Strains)and conventional IPV (Inactivated Poliomyelitis Vaccine Made from Wild Polio Strains) were assign to different group of sequential immunization schedules.

The detail of each group as following:

1)1-dose cIPV + 2-doses bOPV (Candy); 2)1-dose sIPV + 2-doses bOPV (Candy); 3)2-doses cIPV + 1-dose bOPV (Candy); 4)2-doses sIPV + 1-dose bOPV (Candy); 5)2-doses cIPV + 1-dose tOPV (Candy); 6)2-doses sIPV + 1-dose tOPV (Candy); 7)1-dose cIPV + 2-doses bOPV (Liquid); 8)1-dose sIPV + 2-doses bOPV (Liquid); 9)2-doses cIPV + 1-dose bOPV (Liquid); 10)2-doses sIPV + 1-dose bOPV (Liquid); 11)2-doses cIPV + 1-dose tOPV (Liquid); 12)2-doses sIPV + 1-dose tOPV (Liquid).

Blood Sample was collected before vaccination and 28 days after the third dose of vaccination. Neutralization antibody against type I, Type I and Type III poliomyelitis virus were detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The safety of different sequential schedule immunization for the vaccines also been monitored.

The first 10% of subjects in each research site，fecal samples were collected to test polio virus shedding.The 7 times are before the second dose immunization and the 7、14、28 days after the second and the third dose immunization.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (37-42 weeks), birth weight meets the standards (over 2500g), aged from 60 days to 90 days old;
* parent(s) or guardians are able to understand and sign informed consent for participation;
* Participants or guardians are able to attend all planned clinical appointment and obey and follow all study instructions;
* subject didn't administrate with any immunoglobulin after birth (except the Hepatitis B specific immunoglobulin) and did not administrate any other live vaccines within 28 days or inactivated vaccines within 14 days;
* Axillary temperature ≤37.1℃.

Exclusion Criteria:

Subjects will not be eligible for the study if any of the following criteria is met：

* Subject who has a medical histroy with Hypersensitiveness, eclampsia, epilepsy, cerebropathia and neurological illness
* Subject who is allergy to Streptomycin, neomycin and polymyxin B
* Subject with immunodeficency or are in the process of immunosuppressor therapy
* Clinical diagnosis of poliomyelitis;
* Acute febrile disease or infectious disease;
* Labor abnormal, asphyxiation rescues, congenital abnormality, developmental disability, serious chronic diseases;
* Allergic to any ingredient of vaccine or with allergy history to any vaccine;
* Taking orally injecting of steroid hormone over 14 days in the recent month;
* Febrile (temperature ≥ 38.0°C) in three days;
* Diarrhea with one week (more than 3 motions a day);
* Taking part in another clinical trail;
* Any OPV vaccination contraindication and any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Antibody titers of anti-poliovirus antibodies in serum of children who received 2 -doses cIPV/sIPV+1 dose tOPV or 2-doses cIPV/sIPV +1 dose bOPV. | at the 28 days after finishing the 3rd dose
  Based on neutralization test to measure the production of serum antibody. In order to identify what kind of immune programme for children is best. The study will compare the antibody seroconversion rate and antibody geometric mean titers(GMTs) for Type I, Type II and Type III Poliomyelitis after sequential immunization of 2-doses cIPV/sIPV + 1-dose tOPV (Liquid / candy) with 2-doses cIPV /sIPV+ 1-dose bOPV (Liquid/ candy).

SECONDARY OUTCOMES:
Safety:number of adverse events and serious adverse events | within 28 days after each dose injection
  Local and systemic adverse events were active collected and recorded to calculate the number of adverse events and serious adverse events when the subject received each dose of vaccine ，especially the bOPV.
Long term Safety:number of serious adverse events | Up to 6month after finishing the 3rd dose
  Over a period of 6 months the study observed for the safety of each sequential immunization schedule.Serious adverse events were collected and recorded after finishing the 3rd dose.
Antibody titers of anti-poliovirus antibodies in serum of children who received 1 dose cIPV/sIPV+2 dose bOPV(candy/liquid) or 2 doses cIPV/sIPV+1 dose bOPV | at the 28 days after finishing the 3rd dose
  Based on neutralization test to measure the production of serum antibody. In order to identify what kind of immune programme for children is best. The study will compare the antibody seroconversion rate and antibody geometric mean titers(GMTs) for Type I, Type II and Type III Poliomyelitis after sequential immunization .The antibody seroconversion rate and antibody geometric mean titers for type I, type II and Type III of 1-dose cIPV/sIPV + 2-doses bOPV (Liquid/ candy) with 2-doses cIPV/sIPV + 1-dose bOPV(Liquid / candy) .

OTHER OUTCOMES:
Viral shedding | before the second dose;the 7 days after the second dose;the 14 days after the second dose;the 28 days after the second dose;the 7 days after the third dose;the 14 days after the third dose;the 28 days after the third dose
  The first 10% of subjects in each research site，fecal samples were collected to test poliovirus shedding.
  Whether the fecal sample contain polio virus or other enterovirus,using L20B cell and RD cell to solation and identification of polio virus from subjects' fecal suspension sample.
  PCR and serotypes are used to identify of polio virus types（type I、II、III）. The WHO "polio laboratory manual" and the standard "diagnosis for poliomyelitis(WS 294-2016)" of PRC were used for method reference.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Master, Principal Investigator — Guangxi Province Center for Diseases Control and Prevention
Locations (1):
- Guangxi Provincial Center for Diseases Control and Prevention, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Zhao Y, Yang Z, Li Y, Shi H, Zhao T, Yang X, Li J, Li G, Wang J, Ying Z, Yang J. The impact of different IPV-OPV sequential immunization programs on hepatitis A and hepatitis B vaccine efficacy. Hum Vaccin Immunother. 2022 Dec 31;18(1):2024063. doi: 10.1080/21645515.2021.2024063. Epub 2022 Jan 19. PMID 35044877